CLINICAL TRIAL: NCT03109106
Title: Proposed Procalcitonin Re-Implementation Protocol for Johns Hopkins Bayview Medical Center (JHBMC): A Stewardship Project
Brief Title: Procalcitonin for Stewardship in Respiratory Infections A Stewardship Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00120126
Record Dates: First submitted 2017-03-23; First posted 2017-04-12 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: LRTI
Keywords: MICU; CICU; PCT - Procalcitonin; B·R·A·H·M·S PCT sensitive Kryptor®; Antibiotic initiation; Antibiotic de-escalation

STUDY DESIGN:
Intervention Model Description: Will identify eligible patients and controls prospectively in 2 week alternating blocks. Study candidates enrolled during the intervention blocks will receive PCT-guided therapy. Study candidates enrolled during the control periods will receive standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCT Arm (Experimental): oAntibiotic management includes use of a validated PCT algorithm in addition to clinical judgment, other laboratory values, and microbiological pathogen identification. Subjects will be enrolled and data collected prospectively in 2017.
  Patient records will be reviewed for outcomes data and the patients will receive a phone call for outcomes assessment at 30 days post discharge.
  Interventions: Device: PCT Arm
- Control Group (No Intervention): Patients enrolled during the control blocks will receive antibiotics for respiratory infection at the provider's discretion in keeping with current standards of care. Patient records will be reviewed for outcomes data and the patients will receive a phone call for outcomes assessment at 30 days post discharge.

INTERVENTIONS:
Device: PCT Arm — PCT-guided antibiotic therapy per study protocol
  Other Names: B·R·A·H·M·S PCT sensitive KRYPTOR®
  Arms: PCT Arm

SUMMARY:
Antibiotics are overused in hospitals nationwide, leading to unnecessary drug costs and adverse events. Antibiotic stewardship is now a national and international priority and regulatory authorities are mandating antibiotic stewardship programs in all hospitals. Respiratory infections account for a large percentage of antibiotic overuse. Procalcitonin has been shown to help providers significantly shorten the duration of antibiotic therapy in respiratory infections. As such, this institution seeks to evaluate the impact of PCT-guided antibiotic management on antibiotic use in subjects with acute Lower Respiratory Tract Infection (LRTI) with or without sepsis. Multiple studies have been conducted in Europe and demonstrate the safety of the PCT-guided antibiotic management in pneumonia as well as sepsis. This study will apply PCT-guided therapy to those populations in an all-US study evaluating patient outcomes along with safety and efficacy.

DETAILED DESCRIPTION:
The study will enroll 200 patients in the Procalcitonin (PCT)-guided care cohort and 200 patients in the control cohort, using alternating 2 week time blocks until enrollment targets are reached. Patients during control or non-intervention periods will be prospectively identified and enrolled for the purposes of medical record review and follow up, but will not undergo PCT testing.

Patient Identification/ Recruitment: Intervention Periods

Patients will be identified either by the PI, research assistant, or co-investigator using an Epic system list of patients admitted to a medical service (intensive care unit (ICU) or ward) within the past 48 hours with a diagnosis of respiratory infection and receiving antibiotics for <24 hours, or via referrals from the Emergency Department and admitting teams. Candidate patients will have evidence of an acute lower respiratory tract infection (pneumonia or acute exacerbation of chronic bronchitis) as defined as follows:

o New onset within past 28 days

-At least one respiratory symptom: cough, sputum production, dyspnea, tachypnea, pleuritic chest pain, wheezing

Plus: At least one :

* auscultation abnormality suggestive of pneumonia (rales, ronchi, egophony)
* OR a new consolidation on chest radiology consistent with pneumonia
* OR at least one sign of systemic infection: fever >38.1 or white blood cell (WBC) count >10,000 or <4,000 o AND provider initiating empiric antibiotics The PI or co-investigator will contact the primary provider, if the patient was not referred by the team, and ask permission to approach the patient to discuss study participation. The PI or consenting delegate will then obtain written consent from the patient within 48 hours of antibiotic initiation. Baseline PCT will be added on to admission blood obtained prior to initiation of antibiotics after consent is obtained, Patients will be included if first PCT is performed on blood drawn between 0-24 hours prior to antibiotic initiation.

Serial PCT levels will be obtained and antibiotic decisions guided as follows:

1. Inpatient Non-ICU units (Figure 1) - Med A, Med B, Bridgeview Unit,

   • Antibiotic initiation and de-escalation for patients admitted with moderate severity respiratory infections (CURB-65 = 2-3 pneumonia, chronic obstructive pulmonary disease (COPD) exacerbations), based on a Day 0 value and a Day 2 value (repeat q48 hours up through D7 if previous values are >0.25 ug/L). Withhold antibiotics for initial values <0.1-0.25 (recommend a repeat value 4-6 hours later if antibiotics are held), discontinue antibiotics when PCT drops 80% from the peak value or to an absolute value of <0.25 ug/L. [Not routine care] i. If a patient is planned to discharge from the hospital prior to the 48 hour PCT level, the team may draw the lab early for the purposes of discharge antibiotic decisions, provided the values are drawn at least 6 hours apart.

   ii. Recommend use in conjunction with blood cultures in select patients, universal respiratory viral polymerase chain reaction (PCR) panel, urine Streptococcal and Legionella antigens, and sputum cultures ("the diagnostic bundle" similar to Gelfer 2015 and Branche 2015). [Routine care]
2. Intensive Care Unit (Figure 2) -MICU/Cardiac Intensive Care unit (CICU)/ Progressive Care Unit (PCU)

   • Antibiotic de-escalation for patients with severe sepsis and community acquired pneumonia (CAP)/ hospital-acquired pneumonia (HAP) / ventilator associated pneumonia (VAP)/COPD exacerbations, based on a Day 0 value, with daily follow up levels. Discontinuation recommended for a PCT decrease by ≥80% of peak value over the Day 0 value, or to <0.5 ug/L.[Not routine care] i. Recommend use in conjunction with blood cultures, universal respiratory viral PCR panel, urine Streptococcal and Legionella antigens, and sputum cultures ("the diagnostic bundle" similar to Gelfer 2015 and Branche 2015). [Routine care]
3. Emergency Department (ED): No antibiotic prescribing decisions will be made in the Emergency Department using the PCT-guided algorithm for this study. The ED will only be a site of patient identification, referral, and recruitment as well as lab collection.

Patient Identification/ Recruitment: Control Periods Patients will be identified either by the PI, research assistant, or co-investigator using the same EPIC screening process and inclusion strategy described above. The PI, research assistant, or co-investigator will approach the patient and obtain verbal consent to enroll the patient in the comparison cohort. The study team member will notify the primary provider of the patient's consent, but no PCT will be ordered. The patient will receive antibiotics at the provider's discretion.

Physicians overrides will be considered algorithm-compliant if during the initial prescribing decision any of the following conditions exist:

* Respiratory or hemodynamic instability
* Life-threatening comorbidity
* Initial ICU admission
* PCT < 0.1 μg/l: CAP with pneumonia severity index (PSI) V or (Confusion, uremia, respiratory, blood pressure (CURB) 65 >3, COPD with Global Initiative for Chronic Obstructive Lung Disease (GOLD) Class IV
* PCT < 0.25 μg/l: CAP with PSI ≥IV or CURB 65>2, COPD with GOLD Class > III

Physicians may deviate from the algorithm at any point, but deviations for other reasons will be considered "provider discretion." In case of overruling or deviation, a repeated PCT measurement and early discontinuation of antibiotic therapy after 3, 5,or 7 days will be suggested.

Implementation Strategy

Success of procalcitonin use requires confidence and leadership by the physician leaders in a given area, support from ancillary staff (nursing) to obtain timely blood draws and cultures, and prompting for algorithm use by clinical pharmacists or the stewardship team. Since procalcitonin has already been in use at JHBMC for several years, many clinicians are familiar with the test, but are not confident in its utility based on a lack of clinical guidance/ protocol development. The project would require physician champions in each of the service areas in order to educate providers on its use, help distribute the diagnostic algorithms, and encourage implementation. The Antibiotic Stewardship Team is committed to providing needed education and support for all clinical areas, and following up on procalcitonin levels as able.

Antibiotic Stewardship Team:

* To generate pocket cards with PCT algorithms, inclusion, and exclusion criteria (to include Figure 1 + Detailed exclusion criteria on the floor; Figure 2 + detailed exclusion criteria for the ICU).
* To prepare educational materials for providers
* To educate providers on the PCT protocol and evidence for use
* To collect antibiotic use data

Pathology Lab:

• To provide a list of all procalcitonin values to designated person in each unit every day (via secure means).

Physician Lead (2 housestaff, 2 hospitalists, 1 CICU, 1 MICU, 1 PCU):

* To assist with the distribution of algorithms and prompt providers in their service area to use the algorithm.
* To appoint a person to review the PCT results from their unit every day (ideally a Clinical Pharmacy Specialist, or a charge registered nurse (RN), chief resident, etc) and prompt providers to de-escalate antibiotics accordingly.

Timeline for Study:

March 1, 2017- December 30, 2017: Study period

* Algorithm distribution
* Provider education by the Stewardship Team, in coordination with physician lead
* Physician champion-led implementation of daily PCT reviews (at least 5 per day) specific to unit needs and workflow.

  1. Hospitalist service (Bridgeview Unit, Med A, Med B)
  2. House-staff service (Med A, Med B)
  3. ICU services (MICU/ CICU/ PCU)

ELIGIBILITY:
Inclusion Criteria:

* Candidate patients will have evidence of an acute lower respiratory tract infection (pneumonia or acute exacerbation of chronic bronchitis) as defined as follows:

  o NEW onset within past 28 days
* At least one respiratory symptom: cough, sputum production, dyspnea, tachypnea, pleuritic chest pain, wheezing

PLUS: At least one :

* auscultation abnormality suggestive of pneumonia (rales, ronchi, egophony)
* OR a new consolidation on chest radiology consistent with pneumonia
* OR at least one sign of systemic infection: fever >38.1 or WBC >10,000 or <4,000 AND provider initiating empiric antibiotics

Exclusion Criteria:

* - Age <18
* Microbiologically documented infections caused by organisms for which a prolonged duration is standard of care (i.e. Pseudomonas, Acinetobacter, Listeria, Legionella, Pneumocystis, M. tuberculosis, Non-tuberculous mycobacterium (NTM) infection, S. aureus pneumonia or cavitary pneumonia)
* Severe infections due to viruses and parasites with a risk of bacterial translocation (hemorrhagic fever, malaria)
* Infectious conditions requiring prolonged therapy: endocarditis, brain abscess, deep abscess
* Antibiotics already started 24 hours prior to initial PCT value
* Chronic localized infections (i.e. chronic osteomyelitis, mediastinitis, brain abscess)
* Severely immunocompromised patients (HIV with CD4<200, neutropenic with absolute neutrophil count (ANC) <500, patients on immunosuppressive therapy after solid organ transplantation or those with autoimmune disease (corticosteroids allowed but no more than 20 mg/day (prednisone equivalent) for 14 days). Cystic fibrosis
* Active IV drug abuse
* Pregnant patients
* Patients lacking capacity to consent
* Patients admitted for burn injuries
* Patients within 30 days of major intra-thoracic or intra-abdominal surgery
* Patients receiving antibiotics for a non-respiratory infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Antibiotic Exposure | Hospital admission through 30 days post discharge
  Total and median days of antibiotic therapy by subject compared to controls

SECONDARY OUTCOMES:
Length of stay | Hospital admission through 30 days post discharge
  Days of hospitalization of enrolled subjects with acute LRTI receiving antibiotics
Mortality | Hospital admission through 30 days post discharge
  Death from any cause
30-day readmission | 30 days post discharge
  Number of readmissions, stratified by unit
Cost per case | Hospital admission through discharge date, evaluated at 3 months post discharge
  o Total cost of care during hospitalization for each enrolled subjects with suspected LRTI receiving antibiotics. Data will be extracted from hospital charge database.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No